CLINICAL TRIAL: NCT05190887
Title: What do Patients Expect After Scaphoid Fractures?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kuwait Institute for Medical Specialization (Other Government)
Responsible Party: Principal Investigator, Ali Lari, Principle Investigator: Dr Ali Lari - MB BCh BAO, Kuwait Institute for Medical Specialization
Other Study IDs: KuwaitIMS
Record Dates: First submitted 2021-12-04; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Expectations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess patients expectations pre-op and assess their views on their outcome at one year follow up

DETAILED DESCRIPTION:
Using Trauma expectation factor and trauma outcome measure questionnaire. At fracture time and at one year post fracture

Analyse according to age, sex, fracture pattern, type of intervention

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of a scaphoid fracture
* Age > 18
* Consent for one year follow up

Exclusion Criteria:

* Age <18
* Polytrauma (Multiple systems/ Multiple fractures)
* Ipsilateral fractures of the upper limb that may become distracting or affect rehabilitation
* Delayed presentation with higher risk of non-union or avascular necrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with scaphoid fracture
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Patient expectations after scaphoid fractures | 1 Year
  Trauma Expectation Factor (TEF) questionnaire will be used at the time of injury - followed by the Trauma Outcome Measure (TOM) questionnaire at 1 - year post injury. - Together = TEFTOM. A higher TEF score indicates higher expectations of recovery, while a lower indicated poor expectations. Discrepancy between the two scores demonstrate poor correlation between what the patient expects and what the outcome is.

CONTACTS AND LOCATIONS:
Locations (1):
- AlRazi Orthopedic Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided